CLINICAL TRIAL: NCT05350267
Title: Changing Health and Lifestyle Behaviors of Offspring Following Maternal Bariatric Surgery
Acronym: HALO-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: University of Delaware (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2021-0601
Record Dates: First submitted 2022-04-22; First posted 2022-04-28 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Intervention Model Description: Treatment versus enhanced standard of care
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): HALO is a mixed-delivery intervention (online learning, digital technologies, telehealth visits) co-designed with mothers that (a) uniquely tailors intervention content to integrate post-bariatric surgery guidelines to recommendations to reduce child obesity risk, (b) teaches mothers evidence-based parenting behaviors to support intergenerational lifestyle and home food environment changes, and (c) addresses unique barriers to family-level change identified by mothers post-bariatric surgery.
  Interventions: Behavioral: HALO
- Enhanced Standard of Care (Active Comparator): The comparator group will receive monthly mailings of publicly available and age-appropriate handouts on healthy eating, physical activity, screen time, and healthy sleep habits
  Interventions: Behavioral: Enhanced Standard of Care

INTERVENTIONS:
Behavioral: HALO — Health and Lifestyle Behaviors in Offspring, or "HALO" is designed for mothers who recently had bariatric surgery who have a school-aged child. HALO focuses on providing each mother with education and parenting strategies to improve her child's healthy lifestyle behaviors, such as her child's eating and physical activity, while she is engaged in her own lifestyle behavior change after bariatric surgery.
  Arms: Treatment
Behavioral: Enhanced Standard of Care — The comparator group will receive monthly mailings of publicly available and age-appropriate handouts on healthy eating, physical activity, screen time, and healthy sleep habits
  Arms: Enhanced Standard of Care

SUMMARY:
This is the Phase 2 pilot/feasibility randomized controlled trial of HALO (Health And Lifestyle Behaviors In Offspring), a parent-led behavioral intervention targeting a high-risk pediatric population (i.e., residing offspring ages 6-12; body mass index > the 70th and < 120% of the 95th percentiles of mothers with severe obesity) that is uniquely well-timed, when mothers are highly engaged in behavior change and losing weight during the first year following bariatric surgery.

ELIGIBILITY:
Inclusion criteria:

* Female caregivers with a biological child (either sex) aged 6-12 years
* Caregiver is 3-12 months post undergoing a non-device based bariatric surgical procedure
* Caregiver is able to read, write, and speak in English
* Child has a BMI > the 70th and < 120% of the 95th percentile
* Child not currently engaged in weight management (behavioral, pharmacologic)
* Child has no chronic medical conditions or developmental disabilities
* Child resides in her home > 75% of the time
* Child is willing to participate

Exclusion criteria:

* Female caregiver is not pregnant at time of enrollment
* Must not live >75 miles from Cincinnati Children's Hospital Main Campus.
* Child BMI is > 120% of the 95th percentile

Min Age: 6 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2025-03-10 (Actual); Study Completion 2025-03-19 (Actual)

PRIMARY OUTCOMES:
Preliminary Efficacy - Change in child body mass index standardized for age/sex from baseline to 26 weeks (post-treatment) | baseline to 26 weeks (post-treatment)
  Trained assessors will measure child height/weight using a standardized protocol. These measurements will be converted to body mass index (kg/m^2) and then standardized by child age and sex
Preliminary Efficacy - Change in child body mass index standardized for age/sex from baseline to 52 weeks (6-month follow-up) | baseline to 52 weeks (6-month follow-up post-treatment)
  Trained assessors will measure child height/weight using a standardized protocol. These measurements will be converted to body mass index (kg/m^2) and then standardized by child age and sex

SECONDARY OUTCOMES:
Secondary - Change in child daily intake of total kcals, and kcals from red foods, sugar-sweetened beverages, and fruits and vegetables from baseline to 26 weeks (post-treatment) using a 3-day dietary recall | baseline to 26 weeks (post-treatment)
  Child dietary intake (mother-reported) will be assessed by a registered dietician via 3 scheduled 24-hour phone recalls (2 weekdays, 1 weekend) over a 2 week period using a multiple pass method.
Secondary - Change in child daily intake of total kcals, and kcals from red foods, sugar-sweetened beverages, and fruits and vegetables from baseline to 52 weeks (6-month follow-up) using a 3-day dietary recall | baseline to 52 weeks (6-month follow-up post-treatment)
  Child dietary intake (mother-reported) will be assessed by a registered dietician via 3 scheduled 24-hour phone recalls (2 weekdays, 1 weekend) over a 2 week period using a multiple pass method.
Secondary - Change in child minutes of moderate to vigorous physical activity (MVPA) from baseline to 26 weeks (post-treatment) | baseline to 26 weeks (post-treatment)
  Child minutes of moderate to vigorous physical activity will be assessed via a waist-worn actigraph accelerometer for 7 days, with data processed via validated scoring protocols
Secondary - Change in child minutes of moderate to vigorous physical activity (MVPA) from baseline to 52 weeks (6-month follow-up) | baseline to 52 weeks (6-month follow-up post-treatment)
  Child minutes of moderate to vigorous physical activity will be assessed via a waist-worn actigraph accelerometer for 7 days, with data processed via validated scoring protocols
Secondary - Change in mother-reported child feeding practices of restriction, pressure to eat, perceived responsibility, and monitoring from baseline to 26 weeks (post-treatment) | baseline to 26 weeks (post-treatment)
  Mothers will complete the Child Feeding Questionaire with validated scale scores in the areas of restriction, pressure to eat, perceived responsibility, and monitoring. Items are rated on a 5-point Likert scale, with subscales scored as the average. Higher scores indicate greater use of each feeding strategy.
Secondary - Change in mother-reported child feeding practices of restriction, pressure to eat, perceived responsibility, and monitoring from baseline to 52 weeks (6-month follow-up) | baseline to 52 weeks (6-month follow-up post-treatment)
  Mothers will complete the Child Feeding Questionaire with validated scale scores in the areas of restriction, pressure to eat, perceived responsibility, and monitoring. Items are rated on a 5-point Likert scale, with subscales scored as the average. Higher scores indicate greater use of each feeding strategy.
Secondary - Change in child hours of screen time from baseline to 26 weeks (post-treatment) | baseline to 26 weeks (post-treatment)
  Mother-report of her child's leisure-time spent on a "typical week-day" using 3 types of screens (TV, computer/video-games, internet/electronic media).
Secondary - Change in child hours of screen time from baseline to 52 weeks (6-month follow-up) | baseline to 52 weeks (6-month follow-up post-treatment)
  Mother-report of her child's leisure-time spent on a "typical week-day" using 3 types of screens (TV, computer/video-games, internet/electronic media).
Secondary - Change in physical home food environment total kcals, and kcals from sugar-sweetened beverages, snack foods, fruits, and vegetables from baseline to 26 weeks (post-treatment) | baseline to 26 weeks (post-treatment)
  Trained assessors will conduct an open home food inventory. Assessors record the presence of food or beverage items (size and quantity) located in the kitchen and secondary food storage areas (e.g., pantry, basement refrigerator). Foods/beverages without indication of size on packaging will be weighed. Full package size for partially consumed items will be recorded.
Secondary - Change in physical home food environment total kcals, and kcals from sugar-sweetened beverages, snack foods, fruits, and vegetables from baseline to 52 weeks (6-month follow-up) | baseline to 52 weeks (6-month follow-up post-treatment)
  Trained assessors will conduct an open home food inventory. Assessors record the presence of food or beverage items (size and quantity) located in the kitchen and secondary food storage areas (e.g., pantry, basement refrigerator). Foods/beverages without indication of size on packaging will be weighed. Full package size for partially consumed items will be recorded.
Secondary - Change in mother use of encouragement/modeling from baseline to 26 weeks (post-treatment) | baseline to 26 weeks (post-treatment)
  Scale from the Neighborhood Impact on Kids Study will be used to assess 7 healthful eating behaviors (i.e., fruits, vegetables, low-fat snacks). Each item is rated on a Likert scale from 1 (never) to 5 (always), with the average taken across the 7 items. Higher scores mean more healthful modeling.
Secondary - Change in mother use of encouragement/modeling from baseline to 52 weeks (6-month follow-up) | baseline to 52 weeks (6-month follow-up post-treatment)
  Scale from the Neighborhood Impact on Kids Study will be used to assess 7 healthful eating behaviors (i.e., fruits, vegetables, low-fat snacks). Each item is rated on a Likert scale from 1 (never) to 5 (always), with the average taken across the 7 items. Higher scores mean more healthful modeling.

OTHER OUTCOMES:
Change in maternal percent weight loss and body mass index from baseline to 26 weeks (post-treatment) | baseline to 26 weeks (post-treatment)
  Trained assessors will measure mothers' weight and height using a standardized protocol which will be used to calculate maternal percent weight loss and body mass index (kg/m^2).
Change in maternal percent weight loss and body mass index from baseline to 52 weeks (6-month follow-up) | baseline to 52 weeks (6-month follow-up post-treatment)
  Trained assessors will measure mothers' weight and height using a standardized protocol which will be used to calculate maternal percent weight loss and body mass index (kg/m^2).
Change in maternal total kcals from baseline to 26 weeks (post-treatment) using a 3-day dietary recall | baseline to 26 weeks (post-treatment)
  Mother-reported dietary intake will be assessed by a registered dietician via 3 scheduled 24-hour phone recalls (2 weekdays and 1 weekend) over a 2-week period using the multiple-pass method to measure total kcals.
Change in maternal total kcals from baseline to 52 weeks (6-month follow-up) using a 3-day dietary recall | baseline to 52 weeks (6-month follow-up post-treatment)
  Mother-reported dietary intake will be assessed by a registered dietician via 3 scheduled 24-hour phone recalls (2 weekdays and 1 weekend) over a 2-week period using the multiple-pass method to measure total kcals.
Change in mother's minutes of moderate to vigorous physical activity from baseline to 26 weeks (post-treatment) | baseline to 26 weeks (post-treatment)
  Mother minutes of moderate to vigorous physical activity will be assessed via a waist-worn actigraph accelerometer for 7 days, with data processed via validated scoring protocols.
Change in mother's minutes of moderate to vigorous physical activity from baseline to 52 weeks (6-month follow-up) | baseline to 52 weeks (6-month follow-up post-treatment)
  Mother minutes of moderate to vigorous physical activity will be assessed via a waist-worn actigraph accelerometer for 7 days, with data processed via validated scoring protocols.
Change in child emotional functioning from baseline to 26 weeks (post-treatment) using Sizing Me Up | baseline to 26 weeks (post-treatment)
  Sizing Me Up is a child-reported weight-related quality of life measure validated for youth (ages 5-13) that assesses a child's thoughts and experiences in context of his/her "size". Lowered scores on the 4-item child emotional functioning subscale (how their size makes them feel [mad, sad, worried, and frustrated]) will be monitored. Raw scores will be transformed to a 0-100 scale, with higher scores representing better emotional functioning.
Change in child emotional functioning from baseline to 52 weeks (6-month follow-up) using Sizing Me Up | baseline to 52 weeks (6-month follow-up post-treatment)
  Sizing Me Up is a child-reported weight-related quality of life measure validated for youth (ages 5-13) that assesses a child's thoughts and experiences in context of his/her "size". Lowered scores on the 4-item child emotional functioning subscale (how their size makes them feel [mad, sad, worried, and frustrated]) will be monitored. Raw scores will be transformed to a 0-100 scale, with higher scores representing better emotional functioning.
Attendance/Participation rates | baseline to 26 weeks (post-treatment) and 52 weeks (6-month follow-up)
  Thresholds will be used as guides to evaluate whether study achieved goals (e.g., percent) for enrollment (at least 85 percent eligible approached), representativeness (at least 30 percent Non-White), retention (at least 80 percent mother/child dyads in treatment group complete 16-week intervention), and data completion (at least 80 percent complete all 3 assessements).
Implementation - Fidelity | baseline to 26 weeks (post-treatment)
  Thresholds will be used as guides to evaluate whether treatment arm delivered as intended. Fidelity checklists created specifically for each intervention session based on intervention manual.
Implementation - Usability/Satisfaction | baseline to 26 weeks (post-treatment)
  Thresholds will be used a guides to evaluate whether treatment arm mothers' ratings of content accessibility, acceptability, usability, and satisfaction of the HALO program via Likert ratings (Scale 1-5) with higher scores indicating greater usability and satisfaction. Thresholds are mean/item ratings greater than or equal to 4.
Time needed for intervention | baseline to 26 weeks (post-treatment)
  For the treatment arm. time will be assessed in three ways. Time stamp of time watching sessions videos will be recorded. Treatment sessions will be timed to determine average length of time needed. Number of weeks to complete all sessions will be tracked to determine the average length of time needed to execute intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret H Zeller, PhD, Principal Investigator — Cincinnati Chidren's Hospital Medical Center
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Prior to sharing, all data will be de-identified in a HIPAA-compliant fashion. Data sets will be carefully reviewed to make sure that information such as age and sex cannot be used to gather additional information that could potentially identify individual subjects. All categorical demographic variables will be collapsed into categories large enough so that combinations of demographic categories for age, sex, geographic location, etc., will have 10 or more individuals in each cell. All modalities of data will be shared, including raw and aggregate data. Descriptors for all variables shared will be included to prevent misuse or confusion. Any analytical methods utilized to assess the data will be defined in shared formats.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: 12 months following completion of the study
Access Criteria: PI will provide information

DOCUMENTS (1):
  • Informed Consent Form (2024-01-04): https://cdn.clinicaltrials.gov/large-docs/67/NCT05350267/ICF_000.pdf